CLINICAL TRIAL: NCT07269457
Title: Vitamin D3 for Moderate to Mild Traumatic Brain Injury: A Randomized Trial on Inflammation and Recovery (VIMOT)
Acronym: VIMOT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lagos State University (Other)
Collaborators: Lagos State University Teaching Hospital (LASUTH) (Unknown)
Responsible Party: Principal Investigator, Olufemi Idowu, Principal Investigator,, Lagos State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NHREC/LASUCOM-HREC/5/5/25
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Traumatic Brain Injury (TBI) Patients; Neuroinflammation
Keywords: Traumatic Brain Injury (TBI); Neuroinflammation; Vitamin D3; Glasgow Outcome Scale - Extended (GOS-E); Modified Rankin Scale (mRS); Sub-Saharan Africa
MeSH Terms: conditions — Brain Injuries, Traumatic; Neuroinflammatory Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: This study adopts a Phase II, four-arm, parallel-group, randomized, quadruple-blinded, placebo-controlled interventional model designed to evaluate the efficacy and safety of high-dose versus standard-dose vitamin D₃ supplementation in adults with mild-to-moderate traumatic brain injury (TBI). Participants will be stratified by baseline vitamin D status (deficient or sufficient) and randomized into one of four parallel treatment arms. Each group will receive its assigned intervention for three weeks, followed by a 24-week follow-up period. Randomization will be computer-generated using permuted block design to ensure balance, and allocation will be concealed through sequentially numbered opaque envelopes. Blinding will include participants, caregivers, investigators, and outcome assessors.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group A (Deficient + High-Dose D₃) (Experimental): 40,000 IU loading dose on day 1, followed by 4,000 IU daily for 3 weeks
  Interventions: Drug: Vitamin D3 (Cholecalciferol)
- Group B (Deficient + Standard-Dose D₃) (Active Comparator): 2,000 IU daily for 3 weeks
  Interventions: Drug: Vitamin D3 (Cholecalciferol)
- Group C (Sufficient + Standard-Dose D₃) (Experimental): 2,000 IU daily for 3 weeks
  Interventions: Drug: Vitamin D3 (Cholecalciferol)
- Group D (No Intervention): Sufficient + Placebo

INTERVENTIONS:
Drug: Vitamin D3 (Cholecalciferol) — Participants who are vitamin D deficient (<30 ng/mL) will receive oral cholecalciferol 2,000 IU daily for 3 weeks.
  Arms: Group A (Deficient + High-Dose D₃); Group B (Deficient + Standard-Dose D₃); Group C (Sufficient + Standard-Dose D₃)

SUMMARY:
This study is a Phase II, randomized, quadruple-blinded, placebo-controlled clinical trial designed to test whether vitamin D₃ supplementation can improve recovery after mild-to-moderate traumatic brain injury (TBI) in adults.

Traumatic brain injury often leads to inflammation and poor neurological outcomes, and many patients are vitamin D-deficient. Vitamin D₃ is a safe, widely available supplement that may reduce inflammation and support brain recovery.

A total of 240 adults (18-65 years) with mild-to-moderate TBI will be enrolled at Lagos State University Teaching Hospital, Nigeria. Participants will be assigned to one of four groups:

Group A (Deficient + High-Dose D₃): 40,000 IU loading dose, then 4,000 IU daily for 3 weeks Group B (Deficient + Standard-Dose D₃): 2,000 IU daily for 3 weeks Group C (Sufficient + Standard-Dose D₃): 2,000 IU daily for 3 weeks Group D (Sufficient + Placebo): placebo daily for 3 weeks All groups will be followed for 24 weeks. Blood tests at baseline, week 1, week 2, and week 4 will measure inflammation. Neurological recovery will be assessed at weeks 4, 12, and 24 using the Glasgow Outcome Scale-Extended (GOS-E) and Modified Rankin Scale (mRS).

The main outcomes are changes in inflammatory markers. Secondary outcomes include mortality, functional recovery, hospital stay, safety, and cost-effectiveness.

The results may identify a low-cost, scalable treatment to improve outcomes after TBI, especially in low-resource settings.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a leading cause of death and disability globally, with the majority of cases occurring in low- and middle-income countries (LMICs). Secondary brain injury, driven by inflammation, oxidative stress, and neurovascular disruption, is a major determinant of long-term disability. Despite this burden, there are no approved pharmacological therapies targeting the secondary injury cascade. Vitamin D₃ (cholecalciferol), a fat-soluble secosteroid hormone precursor, has immunomodulatory and neuroprotective properties, including suppression of pro-inflammatory cytokines (e.g., TNF-α, IL-6), enhancement of antioxidant defenses, and stabilization of the blood-brain barrier. However, its therapeutic potential in TBI has not been evaluated in randomized trials in LMICs.

This Phase II, four-arm, randomized, quadruple-blinded, placebo-controlled trial will evaluate the efficacy and safety of vitamin D₃ supplementation in adults (18-65 years) with mild-to-moderate TBI. A total of 240 participants will be stratified by vitamin D status at baseline and allocated into one of four groups:

Group A (Deficient + High-Dose D₃): 50,000 IU loading dose on day 1, followed by 4,000 IU daily for 3 weeks.

Group B (Deficient + Standard-Dose D₃): 2,000 IU daily for 3 weeks.

Group C (Sufficient + Standard-Dose D₃): 2,000 IU daily for 3 weeks.

Group D (Sufficient + Placebo): placebo daily for 3 weeks.

The intervention period is 3 weeks, with follow-up to 24 weeks. Randomization will use stratified block design (age, sex, GCS), and blinding will apply to participants, care providers, investigators, and outcome assessors.

Primary endpoints are changes in inflammatory biomarkers (CRP, ESR, SIRI, SII, PLR, NLR) and functional outcomes measured by the Glasgow Outcome Scale-Extended (GOS-E) and Modified Rankin Scale (mRS). Secondary endpoints include all-cause mortality at 28 days and 24 weeks, hospital length of stay, adverse events (e.g., hypercalcemia), and cost-effectiveness expressed as incremental cost-effectiveness ratios (ICERs) per DALY and QALY averted.

Safety monitoring will include weekly serum calcium and renal function tests during supplementation, adverse event documentation, and oversight by an independent Data Safety Monitoring Board (DSMB). The study will be conducted under Good Clinical Practice (GCP) standards, with regulatory approval and institutional ethics board approval.

This trial is designed to generate context-specific, clinically actionable evidence on whether vitamin D₃ supplementation improves recovery following TBI. If effective, the intervention is highly scalable given its low cost, wide availability, and favorable safety profile, with potential integration into national TBI management guidelines in LMICs.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years
* Diagnosed with mild-to-moderate TBI defined by GCS 9-15
* Presenting within 24 hours of head injury
* Willing and able to provide informed consent or have a legal representative provide consent
* Confirmed vitamin D-deficient status (<30 ng/mL) for randomization into treatment arms OR Vitamin D-sufficient (≥30 ng/mL) to be eligible for inclusion in the observational control arm.

Exclusion Criteria:

* Severe TBI (GCS ≤8)
* Prior use of vitamin D supplements within the past month
* History of hypercalcemia or hyperparathyroidism
* Pregnancy or lactation
* Use of immunosuppressive agents (e.g., corticosteroids, cytotoxic drugs)
* Chronic liver disease
* End-stage renal disease
* Any terminal illness or comorbidity with expected survival <3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in C-reactive protein (CRP) | 4 weeks
  Serum levels of CRP in all patients will be measured at baseline, Weeks 1, 2, and 4. The primary analysis will assess the mean percentage reduction in markers between baseline and Week 4 across study arms.

SECONDARY OUTCOMES:
Change in inflammatory biomarkers (ESR, SIRI, SII, PLR, NLR) | 4 weeks
  Serum levels of ESR, SIRI, SII, PLR, NLR in all patients will be measured at baseline, Weeks 1, 2, and 4. The primary analysis will assess the mean percentage reduction in markers between baseline and Week 4 across study arms.
Neurological functional recovery assessed by Glasgow Outcome Scale-Extended (GOS-E) | Week 4, Week 12, and Week 24
  All patients, functional outcome will be measured using structured GOS-E interviews, scored by blinded assessors. Improvement defined as ≥1 category increase from baseline
Neurological functional recovery assessed by Modified Rankin Scale (mRS) | Baseline, Week 4, Week 12, and Week 24
  Disability level of all patients will be assessed with the Rankin Focused Assessment method for mRS. Improvement defined as ≥1 grade reduction compared to baseline

IPD SHARING:
Plan to Share IPD: Yes
The following de-identified individual participant data (IPD) will be shared:
  Baseline demographics (age, sex, socioeconomic status, education level). Clinical characteristics at admission (Glasgow Coma Scale score, time from injury to presentation, comorbidities).
  Laboratory results (serum 25(OH)D levels, calcium, creatinine, CRP, ESR, and other inflammatory markers such as SIRI, SII, PLR, NLR).
  Intervention assignment (treatment arm) and dosing adherence. Neurological outcome measures (Glasgow Outcome Scale-Extended [GOS-E], Modified Rankin Scale [mRS]) at Weeks 4, 12, and 24.
  Clinical outcomes (length of hospital stay, complications, 28-day mortality, 12-week mortality).
  Adverse events and serious adverse events, including severity and relatedness to intervention.
  Cost-related outcomes (hospitalization cost, laboratory investigations, and other direct medical costs).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting information will be available starting 6 months after publication of the primary manuscript and will remain available for 5 years
Access Criteria: Qualified investigators engaged in scientific research with a methodologically sound proposal. De-identified individual participant data, study protocol, statistical analysis plan, and analytic code. Requests should be submitted via email to the Principal Investigator (PI). Upon approval of a data use agreement, data will be transferred securely.